CLINICAL TRIAL: NCT02735473
Title: Choline Supplementation as a Neurodevelopmental Intervention in Fetal Alcohol Spectrum Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSYCH-2016-23989; R01AA024123 (NIH)
Record Dates: First submitted 2016-04-02; First posted 2016-04-12 (Estimated); Results first posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Fetal Alcohol Spectrum Disorders
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders | interventions — Choline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Choline bitartrate (Experimental): Powdered drink mix containing choline bitartrate 19 mg. per kg.
  Interventions: Drug: Choline bitartrate
- Placebo (Placebo Comparator): Powdered drink mix containing matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Choline bitartrate
  Arms: Choline bitartrate
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled trial of choline supplementation in children with Fetal Alcohol Spectrum Disorders (FASD). The primary outcome measures are cognitive measures.

DETAILED DESCRIPTION:
This project is the third in a series of randomized, double-blind placebo-controlled trials of choline bitartrate in children ages 2-5 who have been diagnosed with Fetal Alcohol Spectrum Disorders (FASD). Pre-clinical data suggests that choline may attenuate the cognitive deficits caused by prenatal alcohol exposure (especially memory deficits). This study will evaluate the effects of daily choline supplementation vs. placebo for 9 months. Outcome measures include an elicited imitation memory paradigm, global cognitive functioning, and aspects of executive functioning. The study will also continue to collect safety and tolerability data.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 2 years to 5 years of age
2. Available parent or legal guardian capable of giving informed consent for participation.
3. Documented prenatal alcohol exposure (self-report, social service records, or adoption records).
4. Modified Institute of Medicine (IOM) criteria for Fetal Alcohol Syndrome (FAS), Partial Fetal Alcohol Syndrome (PFAS), or Alcohol-Related Neurodevelopmental Disorder (ARND) (Hoyme, May, et al., 2005).

Exclusion Criteria:

1. Known history of a neurological condition (ex. epilepsy, traumatic brain injury)
2. Known history of a medical condition known to affect brain function.
3. Known history of other neurodevelopmental disorder (ex. autism, Down syndrome)
4. Known history of very low birthweight (<1500 grams)

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R Wozniak, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wozniak JR, Eckerle JK, Gimbel BA, Ernst AM, Anthony ME, Tuominen KA, de Water E, Zeisel SH, Georgieff MK. Choline enhances elicited imitation memory performance in preschool children with prenatal alcohol exposure: a cumulative report of 3 randomized controlled trials. Am J Clin Nutr. 2025 Apr;121(4):921-931. doi: 10.1016/j.ajcnut.2025.02.009. Epub 2025 Feb 14. PMID 39956364

RESULTS

PARTICIPANT FLOW:
Groups:
- Choline Bitartrate: Powdered drink mix containing choline bitartrate 19 mg. per kg.
  Choline bitartrate
- Placebo: Powdered drink mix containing matching placebo
  Placebo
Period: Overall Study
Arm/Group | Choline Bitartrate | Placebo
Started | 23 | 23
Completed | 17 | 16
Not Completed | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Choline Bitartrate | Placebo | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 16 | 33
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 10 | 8 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 0 | 5
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 5 | 7 | 12
  More than one race | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Elicited Imitation Memory Task - Short Delay Memory Measure: 6 Months
Description: Elicited Imitation memory paradigm - short delay memory measure at 6 months; scores are in percentage correct.
Time Frame: Change from baseline to 6 months in percentage correct
Measure: Mean (Standard Deviation); unit: change in percentage correct
Arm/Group | Choline Bitartrate | Placebo
Number analyzed (Participants) | 17 | 16
change in percentage correct | 0.252 (0.578) | 0.183 (0.213)

2. Primary Outcome: Elicited Imitation Memory Task - Short Delay Memory Measure: 9 Months
Description: Elicited Imitation memory paradigm - short delay memory measure at 9 months
Time Frame: Change from baseline to 9 months
Measure: Mean (Standard Deviation); unit: change in percentage correct
Arm/Group | Choline Bitartrate | Placebo
Number analyzed (Participants) | 17 | 16
change in percentage correct | 0.318 (0.126) | 0.668 (0.372)

3. Secondary Outcome: Stanford-Binet Intelligence Scales: 9 Months
Description: Stanford-Binet Intelligence Scales at 9 months; scores are standardized scores (mean 100 points, standard deviation of 15 points)
Time Frame: Change from baseline to 9 months in IQ points
Measure: Mean (Standard Deviation); unit: Percentage change in full-scale IQ point
Arm/Group | Choline Bitartrate | Placebo
Number analyzed (Participants) | 16 | 16
Percentage change in full-scale IQ point | 0.198 (0.175) | 0.008 (0.172)

4. Secondary Outcome: Minnesota Executive Function Scale: 6 Months
Description: Minnesota Executive Function Scale - Early Childhood Version at 6 months
Time Frame: Change from baseline to 6 months
Population: This measure was not collected at the 6-month visit but was completed at the 9-month visit.
Arm/Group | Choline Bitartrate | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Minnesota Executive Function Scale: 9 Months
Description: Minnesota Executive Function Scale - Early Childhood Version at 9 months; scores are in t-scores (mean=50, standard deviation=10)
Time Frame: Change from baseline to 9 months in t-score points
Measure: Mean (Standard Deviation); unit: Percentage change in overall score
Arm/Group | Choline Bitartrate | Placebo
Number analyzed (Participants) | 16 | 14
Percentage change in overall score | 0.007 (0.091) | 0.017 (0.177)

6. Secondary Outcome: NIH Toolbox Flanker Task: 9 Months
Description: NIH Toolbox Flanker Inhibitory and Control Task at 9 months; scores are fully-corrected t-scores (mean=40, standard deviation=10)
Time Frame: Change from baseline to 9 months in fully-corrected t-score points
Measure: Mean (Standard Deviation); unit: Percentage change in fully-corrected t-s
Arm/Group | Choline Bitartrate | Placebo
Number analyzed (Participants) | 13 | 11
Percentage change in fully-corrected t-s | 0.091 (0.372) | -0.169 (0.641)

7. Secondary Outcome: NIH Toolbox Flanker Task: 6 Months
Description: NIH Toolbox Flanker Inhibitory and Control Task at 6 months
Time Frame: Change from baseline to 6 months
Population: This measure was not collected at the 6-month visit. It was, however, collected at the 9-month visit.
Arm/Group | Choline Bitartrate | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Child Behavior Checklist: 6 Months
Description: Child Behavior Checklist - parent report instrument at 6 months
Time Frame: Change from baseline to 6 months
Population: This measure was not collected at the 6-month visit. It was collected at the 9-month visit.
Arm/Group | Choline Bitartrate | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Child Behavior Checklist: 9 Months
Description: Child Behavior Checklist - parent report instrument at 9 months; scores are t-scores (mean=50, standard deviation=10)
Time Frame: Change from baseline to 9 months in t-score points
Measure: Mean (Standard Deviation); unit: Change from baseline in t-score points
Arm/Group | Choline Bitartrate | Placebo
Number analyzed (Participants) | 14 | 16
Change from baseline in t-score points | -1.9 (8.9) | -1.8 (7.35)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected of the 9 months of the study + 1 additional month post-study
Arm/Group | Choline Bitartrate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 17/23 | 16/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Choline Bitartrate (N=23) | Placebo (N=23)
Fishy body odor (General disorders) | 2 (2) | 1 (1)
Hyper/hypo-activity (General disorders) | 7 (11) | 7 (8)
Mood Changed (Psychiatric disorders) | 4 (9) | 7 (8)
Headaches (General disorders) | 1 (1) | 2 (2)
Stomach ache (Gastrointestinal disorders) | 3 (9) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-08): https://cdn.clinicaltrials.gov/large-docs/73/NCT02735473/Prot_SAP_001.pdf
  • Informed Consent Form (2020-01-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT02735473/ICF_000.pdf